## **Cover Letter**

- **Study's Official Title:** Improving the Mobility of Transportation Disadvantaged Older Adults: A Community-Based Intervention for the Hispanic/Latino Population
- Date the Consent Form Created:
  - o Initial Consent Form on June 08th 2020
  - o Most recent consent form on February 22<sup>nd</sup> 2021
- Unique Protocol Identification Number: V. 2020-0391
- NCT Number: It has not been assigned yet.

## **Submitted by:**

Kathy Lee, PhD, LMSW, CDP
Assistant Professor
School of Social Work
University of Texas at Arlington
501 W. Mitchell St. Arlington, TX 76019

kathy.lee@uta.edu

314-971-7258



# The University of Texas at Arlington (UTA)

## **Informed Consent for Studies with Adults**

#### TITLE OF RESEARCH PROJECT

Improving the Mobility of Transportation Disadvantaged Older Adults: A Community-Based Intervention for the Hispanic/Latino Population

#### **RESEARCH TEAM**

Kathy Lee, PhD | School of Social Work | <u>kathy.lee@uta.com</u>
Jessica Cassidy, MSW | School of Social Work | jessica.cassidy@uta.edu

#### IMPORTANT INFORMATION ABOUT THIS RESEARCH PROJECT

The purpose of the study is to gather information on how a new community-based program can help improve adults over the age of 65 to access transportation for health care and daily life activities. This study seeks to understand the transportation habits and health needs of participants to identify existing community resources that best suit each individual's needs. This work was supported by a grant from the Center for Transportation Equity, Decisions and Dollars (CTEDD) funded by U.S. Department of Transportation Research and Innovative Technology Administration (OST-R) and housed at The University of Texas at Arlington. The program in this research provides an opportunity for you to engage with a college student, acted as "a healthy buddy." You will interact with your healthy buddy for two times and share your concerns regarding transportation and health over the phone. Your healthy buddy will identify community-based information and resources that may meet your needs. You will also receive this information via mail. You can choose to participate in this research study if you are (1) over the age 65, (2) not able to drive, (3) a resident in Texas, (4) managing at least one health condition (e.g., diabetes, high blood pressure, etc.), and (5) primarily speaking Spanish.

You might want to participate in this study if you want to meet with someone to learn more about community resources and information regarding transportation and your health needs. However, you might <u>not</u> want to participate in this study if you do not want to talk about your transportation or health needs or if you do not have the time to meet with your health buddy and to answer survey questions.

This study has been reviewed and approved by an Institutional Review Board (IRB). An IRB is an ethics committee that reviews research with the goal of protecting the rights and welfare of human research subjects. Your most important right as a human subject is informed consent. You should take your time to consider the information provided by this form and the research team, and ask questions about anything you do not fully understand before making your decision about participating.

### TIME COMMITMENT

You will expect three calls from us. During the first meeting, you will be asked to complete pre-survey. The second meeting will be made approximately 2-4 weeks from the first meeting. You will spend approximately 1 hour each time (2 hours in total). Then, we will call you after 6 weeks from the second meeting to complete a post-survey. During post-survey, you will be asked to participate in a qualitative interview following the post-survey. The post-survey and the interview will take about 1 hour in total. Follow-up interviews could be conducted, if necessary, to ensure the interpretation of the qualitative data by telephone. A follow-up interview is a possibility and may take about 30 minutes.

IRB Approval Date: 02/22/21

V. 2020-0391.5



# The University of Texas at Arlington (UTA)

## **Informed Consent for Studies with Adults**

### **RESEARCH PROCEDURES**

(1) completing a pre-test survey prior to the program conduct, (2) participating in the Healthy Buddy Program with your healthy buddy, (3) completing a post-test survey after 6 weeks, and (4) completing an in-depth, individual interview after the completion of the project. The survey will be about your demographics, current transportation needs, and computer usage as well as measures of self-efficacy and quality of life. The meetings with your healthy buddy will be set based on your schedule. Research procedures are expected to take place over the phone.

#### **POSSIBLE BENEFITS**

It is unknown whether you will benefit directly from participating in the study. However, the team anticipates that you may benefit from the sessions with your student healthy buddy by knowing community resources and information regarding transportation and your health needs. The broader implications of the proposed research project include improved understanding of the health and transportation challenges faced by Hispanic and Latino older adults. Furthermore, the research may inform the creation of a culturally sensitive and Spanish-language version of the Healthy Buddy Program.

### **POSSIBLE RISKS/DISCOMFORTS**

Overall, the study presents minimal risk. Due to the personalized nature of the program intervention, the assigned interviewer (student healthy buddy) as well as the research team will know your personal information. Some survey and interview questions regarding gender, race and income may cause some discomfort to participants. However, you skip any questions without withdrawing from the study entirely.

#### **COMPENSATION**

You will receive a \$10 Walmart gift card after your participation in a survey prior to the program conduct and a \$15 Walmart gift card after your participation in a survey and an interview after the Healthy Buddy Program ends. The gift card will be mailed to your mailing address within two weeks of your participation each time.

"The Internal Revenue Service (IRS) considers all payments made to research subjects to be taxable income. Your personal information, including your name, address, and social security number, may be acquired from you and provided to UTA's accounting office for the purpose of payment. If your total payments for the year exceed \$600.00, UTA will report this information to the IRS as income and you will receive a Form 1099 at the end of the year. If you receive less than \$600.00 total for payments in a year, you are personally responsible for reporting the payments to the IRS."

### **ALTERNATIVE OPTIONS**

There are no alternative options offered for this study.

### **CONFIDENTIALITY**

The research team is committed to protecting your rights and privacy as a research subject. Dr. Lee is a mandated reporter and certain information (e.g., abuse) cannot remain confidential. However, all paper and electronic data collected from this study will be stored in a secure location on the UTA campus and/or a secure UTA server for at least three (3) years after the end of this research. The individual interview recording will be immediately destroyed after transcription.

The results of this study may be published and/or presented without naming you as a participant. The data collected about you for this study may be used for future research studies that are not described in

IRB Approval Date: 02/22/21

V. 2020-0391.5



# The University of Texas at Arlington (UTA)

## **Informed Consent for Studies with Adults**

this consent form. If that occurs, an IRB would first evaluate the use of any information that is identifiable to you, and confidentiality protection would be maintained.

While absolute confidentiality cannot be guaranteed, the research team will make every effort to protect the confidentiality of your records as described here and to the extent permitted by law. In addition to the research team, the following entities may have access to your records, but only on a need-to-know basis: the U.S. Department of Health and Human Services and the FDA (federal regulating agencies), the reviewing IRB, and sponsors of the study.

#### **CONTACT FOR QUESTIONS**

Questions about this research study or reports regarding an injury or other problem may be directed to Kathy Lee (kathy.lee@uta.edu) if you speak English, Jessica Cassidy (214-997-4442 or <a href="mailto:jessica.cassidy@uta.edu">jessica.cassidy@uta.edu</a>) if you speak Spanish. Any questions you may have about your rights as a research subject or complaints about the research may be directed to the Office of Research Administration; Regulatory Services at 817-272-3723 or <a href="mailto:regulatoryservices@uta.edu">regulatoryservices@uta.edu</a>.

### **CONSENT**

By saying yes, you confirm that you are 65 years of age or older and have understood this information. You have been informed about this study's purpose, procedures, possible benefits and risks. You have been given the opportunity to ask questions before you participate in this study, and you have been told that you can ask other questions at any time. You voluntarily agree to participate in this study. By saying yes, you are not waiving any of your legal rights. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled. You may discontinue participation at any time without penalty or loss of benefits, to which you are otherwise entitled.

| 0 | 0 |
|-----|----|
| Yes | No |

IRB Approval Date: 02/22/21 V. 2020-0391.5